CLINICAL TRIAL: NCT02185027
Title: Observatory of Invasive Procedures and Bleeding in Patients Treated With New Oral Anticoagulants
Acronym: GIHP-NACO
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Floralis (Industry)
Responsible Party: Sponsor
Other Study IDs: DCIC 13 18
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2018-01

CONDITIONS: Venous Thromboembolism; Atrial Fibrillation
Keywords: Oral anticoagulants; Surgery; Haemorrhage; Emergency
MeSH Terms: conditions — Venous Thromboembolism; Atrial Fibrillation; Hemorrhage; Emergencies | interventions — Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- complications and compliance with GIHP recommendations: Description at 1 month post-intervention of an potential event
  Interventions: Other: complications and compliance with GIHP recommendations

INTERVENTIONS:
Other: complications and compliance with GIHP recommendations — Description of complications, compliance, major bleeding events, treatments, reversal strategies.

SUMMARY:
The arrival on the market of direct oral factor Xa and factor IIa inhibitors (dabigatran (Pradaxa®), rivaroxaban (Xarelto®), apixaban (Eliquis®) and others soon to come) raises novel questions among clinicians confronted with the emergency management of patients treated with these new drugs. It is likely that these new oral anticoagulants (NOACs) will eventually win a significant market share in the indications secondary prevention of venous thromboembolism and prevention of cardioembolic events in patients with nonvalvular atrial fibrillation, due to their net clinical benefit and their practicality of use compared with vitamin K antagonists (VKAs).

However, despite the fact that NOACs reduce the incidence of intracranial bleeding by about half compared with VKAs, the risk remains significant; furthermore, in clinical trials, these drugs had little or no effect on reducing the incidence of major extracranial bleeding. In everyday practice, where the indication could be expanded to unselected populations and due to a potential for misuse, it is likely that the incidence of bleeding complications will be higher than that reported in clinical trials. Indeed, the numerous alerts emanating from regulatory agencies in various countries (US, Australia, etc.) bear witness to this, and should serve as a reminder that these anticoagulants have a real potential for bleeding complications and, in the absence of an antidote, there is no validated management strategy.

Furthermore, as these drugs can be prescribed for months or years, patients may eventually be exposed to situations at high hemorrhagic risk, such as emergency surgery or invasive procedures, trauma, etc. Analysis of data from the trial : dabigatran versus warfarin in patients with atrial fibrillation (RE-LY) showed that during the two years of follow-up, approximately 25% of the patients underwent an invasive procedure, ranging from pacemaker insertion to major surgery. Thus, a large proportion of patients treated with NOACs are concerned by this issue.

In anticipation of a gradually increasing influx of patients in a critical situation (active bleeding or need to rapidly secure hemostasis before an invasive procedure), it is urgent to define the conduct to adopt based on the experience gained from the earliest cases. This is the objective of the French-speaking GIHP-NACO observatory set up by the GIHP (French Working Group on Perioperative Hemostasis).

For the moment, then, the management recommendations derive from expert opinions based on pharmacokinetic data and on the partial correction of NOAC-induced hypocoagulability by various nonspecific procoagulants (non-activated or activated prothrombin complex concentrates, recombinant factor VIIa). These procoagulants are currently used in an empirical manner to control bleeding, with as many successes as failures reported in the literature, and their benefit-risk ratio in these patients is therefore uncertain.

DETAILED DESCRIPTION:
The management of critical situations is difficult for several reasons:

* First, there is significant intra- and inter-individual variability in the pharmacokinetics of NOACs, which is further heightened in the critical setting by drug interactions with other agents that interfere with P-GLYCOPROTEIN (P-GP) and cytochrome ( cytochrome P4503A4) in patients who are often elderly and multi medicated, and by rapid variations in renal function, which is essential for elimination of NOACs.
* Second, biological guidance is weak: there is no clearcut therapeutic range nor any validated hemostatic safety cutoff, as is the case with the International Normalized Ratio (INR) for VKAs. Conventional coagulation tests (PT/aPTT) are poorly standardized and difficult to interpret. Assays to measure the serum concentrations of these drugs are not widespread outside of a few teaching hospitals.
* Third, there is a lack of clinical experience. Analyses of critical situations that occurred during clinical trials were done after the fact and the data collected are heterogeneous and incomplete. Clinical cases reported in the literature are rarely well documented.

The objective of the observatory is to rapidly acquire documented and thorough feedback on clinical experience with these new drugs that will be able to confer a higher level of evidence to the management recommendations for treated patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Managed in view of surgery or an invasive procedure, emergency or not
* Managed and hospitalized for active bleeding
* Long-term therapy (in the indication atrial fibrillation or treatment of pulmonary embolism or deep vein thrombosis) by at least one antithrombotic agent from the following list: DABIGATRAN ETEXILATE MESYLATE or RIVAROXABAN or APIXABAN

Exclusion Criteria:

* Pregnant women
* Refusal to participate in the study: listed in the non-inclusion registry
* Antithrombotics indicated for the prevention of venous thromboembolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects managed in view of surgery or an invasive procedure, emergency or not managed and hospitalized for active bleeding with a long-term therapy (in the indication atrial fibrillation or treatment of pulmonary embolism or deep vein thrombosis) by one antithrombotic agent (Dabigatran, Rivaroxaban, Apixaban)
Sampling Method: Non-Probability Sample
Enrollment: 1166 (Actual)
Dates: Start 2013-06; Primary Completion 2016-03 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
complications and compliance with GIHP recommendations | At 1 month
  Association between the incidence rate at 1 month post-intervention of an event among the following complications and compliance with GIHP recommendations (appended) evaluated by a composite endpoint Major cardiovascular event ( acute coronary syndrome, cardiogenic shock, stroke or Transient Ischemic Attack (TIA), Central Nervous System (extra-CNS) thromboembolic event).
  Major bleeding event in the group of patients who had an emergency invasive procedure.
  Continued bleeding after management (treatment, reversal) in the group of patients managed for bleeding.
  Compliance with GIHP recommendations (appended) evaluated by a composite endpoint based on:
  * Observance of reversal strategies
  * Observance of the therapeutic window between the last administration and the procedure, in cases where the NOAC was stopped

SECONDARY OUTCOMES:
NOAC management | during the perioperative period
  All NOAC treatments will be recorded
reversal strategies description | during the perioperative period
  use or not of reversal strategies will be described
Coagulation test results | during the perioperative period
  Coagulation test results will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Albaladejo, MD, Principal Investigator — University Hospital, Grenoble
Locations (41):
- CHU Brugmann, Brussels, Belgium
- France (40):
  - Hôpitaux du Léman, Thonon-les-Bains, haute-Savoie
  - CH Agen, Agen
  - CHU d'Amiens, Amiens
  - CHR Annecy, Annecy
  - CHU Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - CH Castres, Castres
  - CH Chambéry, Chambéry
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CH Alpes leman, Contamine-sur-Arve
  - CHU Dijon, Dijon
  - CH Gap, Gap
  - CHU de Grenoble, Grenoble
  - Groupe Hospitalier Mutualiste Grenoble, Grenoble
  - CHRU Lille, Lille
  - HCL - Edouard Herriot, Lyon
  - HCL - Hôpital de la Croix-Rousse, Lyon
  - HCL - Lyon Sud, Lyon
  - CHU Marseille, Marseille
  - CHU Montpellier, Montpellier
  - Centre Emile Gallé - SINCAL, Nancy
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - CH de Niort, Niort
  - CHU Nimes, Nîmes
  - APHP - Antoine Beclere, Paris
  - APHP - Tenon, Paris
  - APHP Henri Mondor, Paris
  - APHP Hôpital Bichat, Paris
  - APHP Hôpital Cochin, Paris
  - APHP Site St Antoine, Paris
  - Aphp-Hegp, Paris
  - APHP-Hôpital Beaujon, Paris
  - Centre Hôpital Américain, Paris
  - CHU Bicêtre, Paris
  - CHU Rennes, Rennes
  - CHRU Strasbourg - Hôpital Civil, Strasbourg
  - Hôpital d'Instruction des Armées Sainte-Anne, Toulon
  - CHU Toulouse, Toulouse
  - CH Voiron, Voiron

REFERENCES:
- [Background] Pernod G, Albaladejo P, Godier A, Samama CM, Susen S, Gruel Y, Blais N, Fontana P, Cohen A, Llau JV, Rosencher N, Schved JF, de Maistre E, Samama MM, Mismetti P, Sie P; Working Group on Perioperative Haemostasis. Management of major bleeding complications and emergency surgery in patients on long-term treatment with direct oral anticoagulants, thrombin or factor-Xa inhibitors: proposals of the working group on perioperative haemostasis (GIHP) - March 2013. Arch Cardiovasc Dis. 2013 Jun-Jul;106(6-7):382-93. doi: 10.1016/j.acvd.2013.04.009. Epub 2013 Jun 25. PMID 23810130
- [Background] Marlu R, Hodaj E, Paris A, Albaladejo P, Cracowski JL, Pernod G. Effect of non-specific reversal agents on anticoagulant activity of dabigatran and rivaroxaban: a randomised crossover ex vivo study in healthy volunteers. Thromb Haemost. 2012 Aug;108(2):217-24. doi: 10.1160/TH12-03-0179. Epub 2012 May 25. PMID 22627883
- [Background] Sie P, Samama CM, Godier A, Rosencher N, Steib A, Llau JV, Van der Linden P, Pernod G, Lecompte T, Gouin-Thibault I, Albaladejo P; Working Group on Perioperative Haemostasis; French Study Group on Thrombosis and Haemostasis. Surgery and invasive procedures in patients on long-term treatment with direct oral anticoagulants: thrombin or factor-Xa inhibitors. Recommendations of the Working Group on Perioperative Haemostasis and the French Study Group on Thrombosis and Haemostasis. Arch Cardiovasc Dis. 2011 Dec;104(12):669-76. doi: 10.1016/j.acvd.2011.09.001. Epub 2011 Oct 29. PMID 22152517
- [Background] Healey JS, Eikelboom J, Douketis J, Wallentin L, Oldgren J, Yang S, Themeles E, Heidbuchel H, Avezum A, Reilly P, Connolly SJ, Yusuf S, Ezekowitz M; RE-LY Investigators. Periprocedural bleeding and thromboembolic events with dabigatran compared with warfarin: results from the Randomized Evaluation of Long-Term Anticoagulation Therapy (RE-LY) randomized trial. Circulation. 2012 Jul 17;126(3):343-8. doi: 10.1161/CIRCULATIONAHA.111.090464. Epub 2012 Jun 14. PMID 22700854
- [Background] Heidbuchel H, Verhamme P, Alings M, Antz M, Hacke W, Oldgren J, Sinnaeve P, Camm AJ, Kirchhof P; European Heart Rhythm Association. European Heart Rhythm Association Practical Guide on the use of new oral anticoagulants in patients with non-valvular atrial fibrillation. Europace. 2013 May;15(5):625-51. doi: 10.1093/europace/eut083. PMID 23625942
- [Derived] Godon A, Gabin M, Levy JH, Huet O, Chapalain X, David JS, Tacquard C, Sattler L, Minville V, Memier V, Blanie A, Godet T, Leone M, De Maistre E, Gruel Y, Roullet S, Vermorel C, Samama CM, Bosson JL, Albaladejo P; GIHP-NACO Study Group. Management of urgent invasive procedures in patients treated with direct oral anticoagulants: An observational registry analysis. Thromb Res. 2022 Aug;216:106-112. doi: 10.1016/j.thromres.2022.06.005. Epub 2022 Jun 22. PMID 35785621